CLINICAL TRIAL: NCT02416245
Title: Impact of a Beverage Powder Fortified With Multiple Micronutrients (MMN) and Bacopa Monnieri Extract (EBM) on Cognitive Variables in Indian School Children (7-12yrs; Inclusive) After 4 Months of Intervention: a Double Blind, Randomized Controlled Trial
Brief Title: Impact of Beverage Powder With Micronutrients and Brahmi Extract on Cognitive Variables in Indian School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Cambridge Cognition Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 202379
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-06

CONDITIONS: Cognition
MeSH Terms: interventions — Micronutrients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test beverage powder (Experimental): Test beverage powder is fortified with micronutrients and Bacopa monnieri extract. Each sachet contains 32g of treatmemt product and 6g dairy whitener. Entire content of the sachet will be stirred with 180mL of potable lukewarm water, and given orally twice daily
  Interventions: Dietary Supplement: Beverage powder fortified with micronutrients and Bacopa monnieri extract
- Control beverage powder (Placebo Comparator): Control beverage powder is the non-fortified isocaloric powder i.e. without micronutrients and Bacopa Monnieri extract. Each sachet contains 32g of placebo product and 6g dairy whitener. Entire content of the sachet will be stirred with 180mL of potable lukewarm water, and given orally twice daily
  Interventions: Other: Non fortified isocaloric control (without added micronutrients and Bacopa monnieri extract)

INTERVENTIONS:
Dietary Supplement: Beverage powder fortified with micronutrients and Bacopa monnieri extract — Test beverage powder is fortified with micronutrients and Bacopa monnieri extract. Each sachet contains 32g of treatmemt product and 6g dairy whitener. Entire content of the sachet will be stirred with 180mL of potable lukewarm water, and given orally twice daily
  Arms: Test beverage powder
Other: Non fortified isocaloric control (without added micronutrients and Bacopa monnieri extract) — Control beverage powder is the non-fortified isocaloric powder i.e. without micronutrients and Bacopa Monnieri extract. Each sachet contains 32g of placebo product and 6g dairy whitener. Entire content of the sachet will be stirred with 180mL of potable lukewarm water, and given orally twice daily
  Arms: Control beverage powder

SUMMARY:
The aim of the current study is to investigate the beneficial impact of 4 month consumption of a beverage powder fortified with Brahmi (Bacopa monnieri) extract and multiple vitamins and minerals on short term memory as assessed using standardised cognitive test battery.

DETAILED DESCRIPTION:
Bacopa monnieri (Brahmi) from Scrophulariaceae family has been traditionally used in India as 'memory tonic'. Brahmi's use as a cognitive enhancer has led to recent research to investigate a broad spectrum of cognitive domains. Additionally, micronutrient deficiency in children can impair cognitive functions, and micronutrient supplementation can help reduce/prevent deficiencies in those at risk. Several studies have been conducted so far which establish the cognition enahncing abilities of Brahmi, with no major side effects. The aim of the current study is to investigate the beneficial impact of 4 month consumption of a beverage powder fortified with Brahmi extract and multiple vitamins and minerals on short term memory as assessed using standardised cognitive test battery.

ELIGIBILITY:
Inclusion Criteria:

* Z-score of Body Mass Index (BMI) for age of >-2 to <-1
* Participant and participant's parents/legally authorized representatives (LAR) understand and are willing, able and likely to comply with all the study procedures
* Participant is in good general health; has no condition that could affect the safety of participant

Exclusion Criteria:

* Child in care: A child who is placed under the control/protection of an agency/organization/institution by the court/government
* Allergy/Intolerance/Hypersensitivity any study ingredient
* Severe anaemia (Hb<8g/dL); Attention Deficit Hyperactivity Disorder; Reading dyslexia or behavioral disorders
* Health condition that could affect food metabolism; any physical or psychiatric illness that could lead to non-completion of study
* Concurrent use of other health food drinks/supplements, within 1 month prior to study start
* Sibling participation in study

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
'Between errors' in CANTAB task 'Spatial working memory' | Baseline to 4 months
  'Spatial working memory' task measures the 'Short term memory' (working memory). In this task, participants search through a series of boxes until they find a blue chip, which they move to the "home" area on right side of screen. They then look for the next blue chip but NOT in same box as before. For each problem, the participant must NOT return to a box they have previously found a blue chip in. Number of boxes is gradually increased from 3 to 8. 'Between errors' is defined as times the participant revisits a box in which a token has previously been found. This is calculated for all trials of four or more tokens only. Scale ranges from 0 to 180 with lower score indicating a better performance.
'Strategy' in CANTAB task 'Spatial working memory' | Baseline to 4 months
  'Spatial working memory' task measures the 'Short term memory' (working memory). In this task, participants search through a series of boxes until they find a blue chip, which they move to the "home" area on right side of screen. They then look for the next blue chip but NOT in same box as before. Number of boxes is gradually increased from 3 to 8. 'Strategy' is defined as number of distinct boxes used by the participant to begin a new search for a token, within the same problem. Scale ranges from 4 to 28 with a lower score indicating a better performance.

SECONDARY OUTCOMES:
'Total errors (adjusted)' in CANTAB task 'Paired associate learning' | Baseline to 4 months
  'Paired associate learning' task measures the 'Episodic memory'. In this task, boxes are displayed on the screen and open up in a randomised order to reveal a number of patterns. The participant must remember which pattern is in which box. The number of patterns gradually increases up to a number of eight but the participant has multiple attempts to remember each location. 'Total errors (adjusted)' is defined as the number of times the participant choose the incorrect box for a stimulus on assessment problems, plus an adjustment for the estimated number of errors they would have made on any problems, attempts and recalls they did not reach. Scale ranges from 0 to 88 with a lower score indicating a better performance.
'Problems solved in minimum moves' in CANTAB task 'Stockings of Cambridge' | Baseline to 4 months
  This task measures 'Executive functioning'. The participant is shown two displays containing 3 colored balls. The displays are presented in such a way that they can easily be perceived as stacks of colored balls held in stockings or socks suspended from a beam. This arrangement makes the 3-D concepts involved apparent to the participant, and fits with the verbal instructions. The participant must use the balls in the lower display to copy the pattern shown in the upper display. The balls may be moved one at a time by touching the required ball, then touching the position to which it should be moved. The time taken to complete the pattern and the number of moves required are taken as measures of the subject's planning ability. 'Problems solved in minimum moves' is defined as the number of occasions upon which the participant has successfully completed a test problem in the minimum possible number of moves. Scale ranges from 0 to 14 with a higher score indicating a better performance.
'A Prime' in CANTAB task 'Rapid Visual Information Processing' | Baseline to 4 months
  'Rapid Visual Information Processing' task measures 'Sustained attention'. In this task, the screen will display a box which randomly flashes the numbers 2-9. The participant must press the button on the screen to respond when they see a target sequence of 3-5-7. 'A Prime' is defined as a signal detection measure of sensitivity to the target, regardless of tresponse tendency. This metric is a measure of how good the participant is at detecting target sequences. Scale ranges from 0 to 1 with a higher score indicating a better performance.
'Median latency' in CANTAB task 'Rapid Visual Information Processing' | Baseline to 4 months
  'Rapid Visual Information Processing' task measures 'Sustained attention'. In this task, the screen will display a box which randomly flashes the numbers 2-9. The participant must press the button on the screen to respond when they see a target sequence of 3-5-7. 'Median latency' is defined as the median response latency during assessed blocks where the participant responds correctly. Scale ranges from 100 to 1900 with a lower score indicating a better performance.
'Total false alarms' in CANTAB task 'Rapid Visual Information Processing' | Baseline to 4 months
  'Rapid Visual Information Processing' task measures 'Sustained attention'. In this task, the screen will display a box which randomly flashes the numbers 2-9. The participant must press the button on the screen to respond when they see a target sequence of 3-5-7. 'Total false alarms' is defined as the number of times the participant responds outside the response window of a target sequence. Scale ranges from 0 to 546 with a lower score indicating a better performance.
CANTAB Score on 'Raven's colored progressive matrices' | Baseline to 4 months
  This is a non verbal visual test, assessing the problem solving and reasoning ability. Participants are presented with 36 visual patterns (with one piece missing from the bottom right corner), grouped in three sets of 12 items each. For each visual pattern, participants are presented with various alternative pieces that could complete the puzzle, and have to choose the correct one. Participants have to attempt all 36 items of the task, the final score being the sum of correct answers across the three series. Scale ranges from 0 to 60 with a higher score indicating a better performance.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pune, India